CLINICAL TRIAL: NCT04507919
Title: Managed Access Program (MAP) Cohort Treatment Plan CTMT212X2002I to Provide Access to Trametinib and Dabrafenib Combination Therapy for Patients With BRAF V600 Mutation-positive Advanced Non-Small Cell Lung Cancer (NSCLC).
Brief Title: Managed Access Program Cohort Treatment Plan CTMT212X2002I to Provide Access to Trametinib and Dabrafenib Combination Therapy for Patients With BRAF V600 Mutation-positive Advanced Non-Small Cell Lung Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212X2002I
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer, lung adenocarcinoma; Squamous cell lung carcinoma; Large-cell lung carcinoma; Non small cell lung carcinoma; Non small cell lung cancer; Non-small cell lung cancer; NSCLC; Large cell lung carcinoma; Large cell lung cancer; Compassionate Use; Cohort; Trametinib; Dabrafenib; TMT212
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — dabrafenib; BID protein, human

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Dabrafenib — 150 mg
  Other Names: twice daily (BID)
Drug: Trametininb — 2.0 mg
  Other Names: once daily (QD)

SUMMARY:
The purpose of this Managed Access Program (MAP) Cohort Treatment Plan is to provide guidance to the Physician for the treatment and monitoring of eligible patients diagnosed with BRAF V600E/K activating mutation-positive advanced NSCLC using trametinib/dabrafenib in the Cohort MAP CTMT212X2002I.

The Physician should follow the suggested treatment guidelines. Furthermore, the Physician must comply with the MAP Agreement Letter and applicable local laws and regulations.

DETAILED DESCRIPTION:
Prior to inclusion of a patient in the Cohort, the requesting Physician must submit a request for access to the product in GEMS (Grants, External Requests and Managed Access System) accessible through https://www.novartis.com/our-focus/healthcare-professionals/managedaccess-programs providing the rationale for the request and relevant medical history of the patient.

The request is then assessed against the MAP and Cohort inclusion/exclusion criteria by the medical team experienced with the product and indication. Upon the required approvals, the patient is included in the Cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Has or is willing to give consent to the Treating Physician in accordance with the local regulatory requirements, with age at the time of consent ≥18 years.
2. Has the following diagnosis: Advanced (inoperable, metastatic or locally advanced, e.g. Stage IIIB, Stage IV) NSCLC (Non-Small Cell Lung Cancer) with confirmed BRAF V600E/K activating mutation.
3. Patient is not eligible for any ongoing clinical trial in the same indication.
4. Is receiving care at a clinical site with a Treating Physician who has experience with administering investigational agents for the end-stage NSCLC population, or the patient is willing and/or able to travel to a site and receive treatment under the guidance of physician with this experience. NOTE: The latter option would require the patient being evaluated in advance by the Treating Physician at the experienced site and his/her agreement to assume responsibility for the care of the patient.
5. Is able to retain oral medication and swallow tablets/capsules (appropriate exceptions allowed for patients who are unable to swallow tablets/capsules - this is subject to availability of alternative (liquid) oral formulations).
6. Does not require treatment with any (other) anti-cancer medication (exceptions might be allowed and are subject to individual evaluation).
7. For patients with active brain metastases: the patient does not require or is ineligible for immediate local treatment.
8. Is not eligible for participation in any ongoing clinical trials with dabrafenib and/or trametinib or has recently completed a clinical trial that has been terminated and, after considering other options (e.g., trial extensions, amendments, etc.), the clinical team has determined that treatment is necessary and there are no other feasible alternatives for the patient.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 3 (or equivalent) and is in stable clinical condition. NOTE: patient in rapidly deteriorating clinical condition prior to start of therapy should not be considered for this program.
10. Does not require treatment with prohibited concomitant medications.
11. Women of childbearing potential must have a serum beta-human chorionic gonadotropin (HCG) pregnancy test performed within 14 days prior to starting dabrafenib and trametinib treatment. Patients with a positive pregnancy test result are not eligible for the program. Patients with a negative pregnancy test result must agree to use an effective contraception method as described below throughout the treatment period and for a total of 16 weeks following the last dose of treatment.

    Contraceptive Methods for Females of Childbearing Potential:

    Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during dosing and for 16 weeks after stopping treatment with trametinib (for trametinib monotherapy trials); 2 weeks after stopping treatment with dabrafenib (for dabrafenib monotherapy trials); 16 weeks after stopping treatment with trametinib or 2 weeks after stopping treatment with dabrafenib whichever is longer (for trials of dabrafenib in combination with trametinib).

    Highly effective contraception methods include: (for dabrafenib monotherapy or combination therapy with trametinib)
    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Sterilization (at least 6 months prior to screening) for male partners. The vasectomized male partner should be the sole partner for that subject.
    * Placement of a hormonal or non-hormonal intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year.

    Notes:

    Double-barrier contraception: condom and occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/cream/suppository) are not considered highly effective methods of contraception.

    Hormonal-based methods (e.g. oral contraceptives) are not considered as highly effective methods of contraception due to potential drug-drug interactions with dabrafenib Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

    If a patient becomes pregnant during the treatment period of the program, the treatments should be stopped immediately.
12. Written patient informed consent must be obtained by the Treating Physician prior to start of treatment in accordance with the applicable local regulatory requirements.

Medical exclusion criteria

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Female who is pregnant or nursing (patient must discontinue nursing in order to enroll in the program).

   NOTE: Safety and efficacy in pregnant or nursing women has not been investigated.

   Inclusion of pregnant or nursing woman may be considered in individually upon review by the Novartis Country Pharma Organization Medical Advisor/Director.
2. Patients who have any lab abnormalities or AE/SAEs greater than Grade 3 (CTCAE v5.0).
3. Concurrent treatment with other systemic anti-cancer therapies is not allowed, with the exception of whole brain radiation and brain radiosurgery. Patients who are currently being treated with another systemic anti-cancer therapy (e.g., chemotherapy, immune, biologic, or targeted therapy) must discontinue use prior to initiation of treatment with trametinib and dabrafenib. NOTE: Radiation skin injury has been reported with concurrent use of dabrafenib and radiation. All AEs/SAEs related to WBRT (whole brain radiation) or brain radiosurgery are required to resolve to Grade 1 or less (CTCAE 5.0) prior to start of the program treatment.
4. Patients who have received prior therapy with a BRAF inhibitor other than dabrafenib.

   NOTE: Consideration may be given to those patients who have either (1) received prior BRAF therapy and there is disease progression in the CNS only or (2) discontinued prior BRAF therapy due to an adverse event that is not likely to recur in response to treatment with Dabrafenib.
5. Presence of malignancy other than NSCLC within 1 year of enrolment into this program or any malignancy with confirmed activating RAS mutation. Patient with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma is eligible. NOTE: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility.
6. Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib or dabrafenib, or excipients or to dimethyl sulfoxide (DMSO).
7. Current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy.
8. Current evidence of cardiovascular risk including any of the following:

   * LVEF<LLN
   * A QT interval corrected for heart rate using the Bazett's formula ≥ 480 msec;
   * Clinically significant uncontrolled arrhythmias
   * Acute coronary syndromes (including myocardial infarction and unstable angina).
   * Congestive heart failure ≥ Class II as defined by New York Heart Association
9. Known history for testing positive for Human Immunodeficiency Virus (HIV).
10. Not able to understand and to comply with treatment instructions and requirements.
11. History of hypersensitivity to any drugs or metabolites of similar chemical classes as the product.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult